CLINICAL TRIAL: NCT07071376
Title: Effect of Cold Dialysis Application on Postdialysis Fatigue in Hemodialysis Patients
Brief Title: Cold Dialysis in Hemodialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Gülay Turgay, assistant professor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dialysis
Record Dates: First submitted 2025-06-16; First posted 2025-07-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dialysis Related Complication
Keywords: dialysis; cold dialysis; fatique

STUDY DESIGN:
Intervention Model Description: Cold dialysis group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold Dialysis (Experimental): To be applied with cold dialysis
  Interventions: Other: cold dialysis

INTERVENTIONS:
Other: cold dialysis — Patients who meet the inclusion criteria will receive 3 sessions of cold dialysis treatment by reducing the dialysate temperature from 36.5°C to 36°C. Patients will receive this treatment for 1 week, i.e. 3 dialysis sessions. Each dialysis session will last 4 hours. During each dialysis session, the thermal comfort status of the patients will be evaluated by applying the Temperature Comfort Perception Scale at the beginning of dialysis, at the 1st, 2nd and 3rd hours of dialysis and at the end of dialysis. In addition, the day after each session, the patients will be called by phone and the Postdialysis Fatigue Scale will be re-administered and their fatigue levels will be evaluated.

SUMMARY:
The standard dialysate temperature is usually set at 36.5°C in hemodialysis applications. Since this temperature is close to the patient's body temperature, it is ideal for preventing the patient from experiencing hypothermia while ensuring cardiovascular stability. In the literature, it is seen that changing the dialysate temperature, especially cold dialysis applications, is used in the management of nausea, the effect on vital signs, determining hemodialysis adequacy and common complications, and in the management of symptoms such as hypotension, cardiac stability, vascular stability, fatigue, and muscle cramps. However, no study has been found using cold dialysis in the management of fatigue that develops after dialysis.Therefore, the aim of this study is to examine the effect of cold dialysis application on post-dialysis fatigue in patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effect of cold dialysis application on post-dialysis fatigue in patients receiving hemodialysis treatment.

Research Hypothesis

H1: Cold dialysis application reduces the level of post-dialysis fatigue.

METHOD

Research Design

This study was designed as a single group pre-test-post-test experimental design.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study
* Age 18 and over
* Having been on hemodialysis for at least 6 months
* Having hemodialysis 3 times a week
* Having a high postdialysis fatigue score cut-off point compared to the mean

Exclusion Criteria:

* Having an active infection
* Having a body temperature above 37.5°C
* Having serious cardiovascular diseases (e.g., uncontrolled hypertension, congestive heart failure)
* Having a history of acute complications during dialysis
* Having a history of severe hypotension
* Patients whose dialysis treatment was interrupted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Post-dialysis fatigue scale | 1 week
  A minimum score of 11 and a maximum score of 55 is obtained from this scale, and an increase in the score indicates an increase in the severity of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Turgay, Study Director — Baskent Universitesi
Locations (1):
- Baskent University, Ankara, Türkiye, Turkey (Türkiye)